CLINICAL TRIAL: NCT00813774
Title: Open, Randomized, Parallel Group, Single Dose, Bioavailability Comparison of 3 Certolizumab Pegol Solution Formulations (Lyophilized, Liquid, Pre-filled Syringe Formulation) to Healthy Volunteers
Brief Title: Bio-availability Comparison of Three Formulations of Certolizumab Pegol in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RA0003; Eudract no. 2007-006344-22
Record Dates: First submitted 2008-12-19; First posted 2008-12-23 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Bioavailability Study on Healthy Volunteers
Keywords: Cimzia; certolizumab pegol; Bioavailability; Healthy volunteers
MeSH Terms: interventions — Certolizumab Pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Reference (Active Comparator): Lyophilized formulation (reference)
  Interventions: Biological: Certolizumab pegol
- Liquid (Experimental): Liquid Formulation (test)
  Interventions: Biological: Certolizumab pegol
- Pre-filled Syringe (Experimental): Pre-filled syringe (test)
  Interventions: Biological: Certolizumab pegol

INTERVENTIONS:
Biological: Certolizumab pegol — Lyophilized certolizumab pegol vial of 200mg for reconstitution of a solution with 1 mL water for injection, single dose of 400 mg given as two subcutaneous injections of 200mg
  Other Names: Cimzia; CDP870
  Arms: Reference
Biological: Certolizumab pegol — Certolizumab pegol liquid formulation 200 mg/mL in 1 mL vial single dose of 400 mg given as two subcutaneous injections of 200mg
  Other Names: Cimzia; CDP870
  Arms: Liquid
Biological: Certolizumab pegol — 200 mg/1 mL liquid certolizumab pegol solution in a pre-filled syringe, single dose of 400 mg given as two subcutaneous injections of 200mg
  Other Names: Cimzia; CDP870
  Arms: Pre-filled Syringe

SUMMARY:
To compare the bioavailability of a single dose of certolizumab pegol solutions given subcutaneously either by one of the three formulations and to investigate safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers aged between 18 and 55
* Body Mass Index (BMI) between 18 and 30 kg/m2 with normal laboratory data
* negative for Tuberculosis test
* normal Electrocardiogram (ECG)
* adequate contraception for females
* given informed consent

Exclusion Criteria:

* Any significant abnormality in medical history, physical examination, laboratory testing
* Intake of concomitant medication
* smoking more than 10 cigarettes per day
* alcohol or drug abuse
* pregnancy or breast feeding
* history of tuberculosis
* participation in another trial within 3 months prior to this study
* previous administration of certolizumab pegol

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 149 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve from time 0 to infinity (AUC) | PK samples: from pre-dose to Week 12
Area under the plasma drug concentration-time curve from time 0 to the last quantifiable point (AUC(0-t),) | PK samples: from pre-dose to Week 12
Maximum plasma concentration (Cmax) | PK samples: from pre-dose to Week 12

SECONDARY OUTCOMES:
Time point where log-linear elimination phase begins (TLIN ) | PK samples: from pre-dose to Week 12
Lowest quantifiable concentration time (LQCT) | PK samples: from pre-dose to Week 12
Apparent terminal elimination rate constant (λz) | PK samples: from pre-dose to Week 12
Apparent terminal elimination half-life (t1/2) | PK samples: from pre-dose to Week 12
Time corresponding to Cmax (tmax) | PK samples: from pre-dose to Week 12
Apparent Total body clearance (CL/F) | PK samples: from pre-dose to Week 12
Apparent Volume of distribution (Vz/F) | PK samples: from pre-dose to Week 12
Extrapolated portion of the AUC (AUC_ext ) | PK samples; from pre-dose to Week 12
Number of subjects with anti-certolizumab pegol antibody plasma level >2.4 units/mL | PK samples; from pre-dose to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (2):
- France (2):
  - Rennes
  - Rueil-Malmaison